CLINICAL TRIAL: NCT04608240
Title: Dose Surgical Pleth Index Play a Role to Predict Optimal Timing for Tracheal Intubation During Anesthetic Induction?
Brief Title: Surgical Pleth Index: Predicting the Optimal Timing for Tracheal Intubation During General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director of the department of anaesthesiology, Shanghai cancer center, Fudan University
Other Study IDs: SPI V 1.0
Record Dates: First submitted 2020-10-02; First posted 2020-10-29 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Trachea Intubation
Keywords: surgical pleth index; hemodynamic reactivity; trachea intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical pleth index (SPI) has been widely investigated in assessing the nociceptive level, and tracheal intubation is a noxious stimulus during the induction of anesthesia. This study aims to evaluate the ability of SPI to predict hemodynamic reactivity after tracheal intubation, and find the target value of SPI to guide the optimal timing for tracheal intubation.

DETAILED DESCRIPTION:
The surgical pleth index (SPI)monitored by a oxygen saturation (Spo2) probe, is a dimensionless score which is based on the photoplethysmographic analysis of the pulse wave and the heartbeat interval. SPI score monitored during surgery is the indicator that may reflect a patient's autonomic response to certain noxious stimulus and is correlated to his/her nociception level. Once noxious stimulus occur, sympathetically-mediated vasoconstriction and cardiac autonomic tone increasing can be reflected by SPI. Several studies have since investigated the potential benefits of SPI-guided anesthesia, such as SPI could reduce the intraoperative opioid consumption and facilitate extubation after surgery.Jain N et al. found that the need for postoperative analgesics decreased although fentanyl consumption increased, when SPI guided opioid use Intraoperatively . The level of SPI was also reported to be able to predict postoperative pain, which could guide clinical use of opioids and improve patient postoperative satisfaction.

Recent studies on SPI mainly focus on the maintenance period of anesthesia and postoperative analgesia, and there is few studies on the application of SPI in anesthesia induction period. Hemodynamic stability in induction period has always been the technical key point that anesthesiologists pay attention to, especially for patients with cardiovascular and cerebrovascular diseases, maintaining hemodynamic stability is particularly important. Endotracheal intubation is a common procedure during general anesthesia. The hemodynamic fluctuation caused by intubation stimulation is usually caused by the premature timing of intubation.

At present, the timing of intubation is much depended on the clinical experience of an anesthesiologist, such as according to the degree of blood pressure, heart rate decline or predicted onset of propofol,opioid and neuromascular blocker. This study aims to explore whether the SPI can be used in quantitative prediction of intubation timing or prediction the hemodynamic reactivity after intubation, and to investigate the influence of age and gender on SPI value.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status (ASA) 1-2
* Patients aged 18-80 years undergoing non-emergency anesthesia

Exclusion Criteria:

* age <18 years
* severe peripheral or cardiac neuropathy
* significant arrhythmia (i.e. atrial fibrillation or atrioventricular block)
* pacemaker
* neurovascular diseases
* uncontrolled hypertension
* treatment with vasoactive medication during the induction of anesthesia
* any intraoperative treatment with beta receptor blockers, clonidine, beta receptor agonists, or any other drug suspected to interact with the sympathovagal balance
* predicted difficult ventilation
* chronic pain requiring long-term analgesics
* addictive to opioids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Society of Anesthesiology physical status (ASA) 1-2 and patients aged 18-80 years undergoing non-emergency anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
ability of SPI to predict hemodynamic reactivity after tracheal intubation in general population | within 2 minutes after trachea intubation
  The area under receiver-operating characteristic curve (AUC) of SPI
ability of SPI to predict hemodynamic reactivity after tracheal intubation in female | within 2 minutes after trachea intubation
  The area under receiver-operating characteristic curve (AUC) of SPI
ability of SPI to predict hemodynamic reactivity after tracheal intubation in male | within 2 minutes after trachea intubation
  The area under receiver-operating characteristic curve (AUC) of SPI

SECONDARY OUTCOMES:
influence factors of hemodynamic reactivity | within 2 minutes after trachea intubation
  using logistic regression model
Cardiovascular stress level | within 2 minutes after trachea intubation
  delta rate pressure product (ΔRPP) between different ranges of SPI

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Department of Anesthesiology, Fudan University Shanghai Cancer Center; Department of Oncology, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Struys MM, Vanpeteghem C, Huiku M, Uutela K, Blyaert NB, Mortier EP. Changes in a surgical stress index in response to standardized pain stimuli during propofol-remifentanil infusion. Br J Anaesth. 2007 Sep;99(3):359-67. doi: 10.1093/bja/aem173. Epub 2007 Jul 3. PMID 17609248
- [Background] Bergmann I, Gohner A, Crozier TA, Hesjedal B, Wiese CH, Popov AF, Bauer M, Hinz JM. Surgical pleth index-guided remifentanil administration reduces remifentanil and propofol consumption and shortens recovery times in outpatient anaesthesia. Br J Anaesth. 2013 Apr;110(4):622-8. doi: 10.1093/bja/aes426. Epub 2012 Dec 5. PMID 23220856